CLINICAL TRIAL: NCT01211821
Title: Effect of BMS-914392 on the Pharmacokinetics of Metoprolol and on Heart Rate After Co-administration of BMS-914392 and Metoprolol in Healthy Subjects
Brief Title: Effect of BMS-914392 on Pharmacokinetics of Metoprolol
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: CV203-003
Record Dates: First submitted 2010-09-03; First posted 2010-09-30 (Estimated); Last update posted 2011-02-02 (Estimated); Status verified 2011-02

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Metoprolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- metoprolol (Other): Treatment A
  Interventions: Drug: metoprolol
- BMS-914392 + metoprolol (Experimental): Treatment B
  Interventions: Drug: metoprolol; Drug: BMS-914392

INTERVENTIONS:
Drug: metoprolol — Tablets, Oral, 200 mg, once, 1 day
Drug: BMS-914392 — Tablets, Oral, 60 mg, once daily, 7 days
  Arms: BMS-914392 + metoprolol

SUMMARY:
The purpose of the study is to assess the effects of BMS-914392 administration on the pharmacokinetics of a single-dose of metoprolol in healthy subjects.

DETAILED DESCRIPTION:
Protocol designed to evaluate the potential for a drug-drug-interaction

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects as determined by no clinically significant deviation from normal in medical history, physical examination, ECGs, and clinical laboratory determinations.
* Subjects genotyped as Intermediate, Extensive or Ultra-rapid CYP2D6 metabolizers
* Women of childbearing potential (WOCBP) and men must be using an acceptable method of contraception to avoid pregnancy

Exclusion Criteria:

* Any significant acute or chronic medical illness.
* Current or recent (within 3 months of study drug administration) gastrointestinal disease.
* Current or history of neurological diseases or psychiatric disorders, cardiovascular diseases, and bronchospastic diseases.
* CYP2D6 poor metabolizers based on genotype

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2010-09; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of single dose of metoprolol derived from serial measurements of metoprolol plasma concentrations | Pre-dose and 0.5 Hr, 1 Hr, 1.5 Hr, 2 Hr, 3 Hr, 4 Hr, 6 Hr, 8 Hr, 12 Hr, 24 Hr, and 36 Hr after dosing of metoprolol alone or in combination with BMS-914392

SECONDARY OUTCOMES:
The effect of multiple doses of BMS-914392 on PR, QRS, RR, and QTc intervals derived from serial electrocardiograms (ECGs) | Pre-dose and 0.5 Hr, 1 Hr, 1.5 Hr, 2 Hr, 3 Hr, 4 Hr , 6 Hr, 8 Hr, 12 Hr, 24 Hr after dosing with metoprolol alone or in combination with BMS-914392
Number of subjects with adverse events as a measure of safety and tolerability of BMS-914392 | Daily

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Pra International, Lenexa, Kansas, United States

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx